CLINICAL TRIAL: NCT03104881
Title: Comparisons of Two Types of Rehabilitation Robot for Upper Extremities: 3 Dimension Exoskeleton Type Upper Extremity Robot vs. 2 Dimension End-effector Type Robot): Randomized Controlled Trial
Brief Title: Comparisons of Two Types of Rehabilitation Robot for Upper Extremities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2015-01-005
Record Dates: First submitted 2016-10-23; First posted 2017-04-07 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3D exoskeleton type robot (Experimental): 3 dimension exoskeleton type upper extremity robot
  Interventions: Device: 3D exoskeleton type robot
- 2D end-effector type robot (Experimental): 2 dimension end-effector type upper extremity robot
  Interventions: Device: 2D end-effector type robot

INTERVENTIONS:
Device: 3D exoskeleton type robot — 3 dimension exoskeleton type upper extremity robot
  Arms: 3D exoskeleton type robot
Device: 2D end-effector type robot — 2 dimension end-effector type upper extremity robot
  Arms: 2D end-effector type robot

SUMMARY:
Comparisons of two types of rehabilitation robot for upper extremities: 3 dimension exoskeleton type upper extremity robot vs. 2 dimension end-effector type robot)

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Onset ≥ 3 months
* 8 ≤ Fugl-Meyer Assessment score ≤ 30
* Shoulder or elbow flexor spasticity modified ashworth scale ≤ 3
* Cognitively intact enough to understand and follow the instructions from the investigator

Exclusion Criteria:

* History of surgery of affected upper limb
* Fracture of affected upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change of Fugl-Meyer Assessment | Fugl-Meyer Assessment change from baseline at 4 weeks
Wolf motor function test | Fugl-Meyer Assessment change from baseline at 4 weeks

SECONDARY OUTCOMES:
Wolf motor function test | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
Motor status score | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
medical research council scale of upper extremity | baseline
Modified Ashworth scale of upeer extremity | baseline
Pain of upper extremity | from baseline to 4 weeks after baseline
  Pain complaints from participants
Stroke impact scale | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
Smoothness | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
  Kinematics from Inmotion2 during point-to-point
Reach Error | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
  Kinematics from Inmotion2 during point-to-point
Path Error | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
  Kinematics from Inmotion2 during point-to-point
Mean velocity | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
  Kinematics from Inmotion2 during point-to-point
Maximum velocity | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
  Kinematics from Inmotion2 during point-to-point
Cricle size | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
  Kinematics from Inmotion2 during circle drawing
Cricle independence | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
  Kinematics from Inmotion2 during circle drawing
Intrinsic motivation inventory | 4 weeks after baseline
stroke rehabilitation motivation scale | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline
Beck depression index | baseline, 4 weeks after baseline, 8 weeks after baseline, 10 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, Seoul, South Korea

REFERENCES:
- See also: Site of the present study — http://nrc.go.kr